CLINICAL TRIAL: NCT00376688
Title: Phase II Trial of CCI-779 (Temsirolimus) in Patients With Locally Advanced or Metastatic Breast Cancer
Brief Title: Temsirolimus in Treating Patients With Locally Advanced or Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02703; NCI-2012-02703 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NCI-7674; UCCRC-14705A; CDR0000495399; UCIRB 14705A; 14705A; 7674 (Other: University of Chicago Comprehensive Cancer Center); 7674 (Other: CTEP); P30CA014599 (NIH); NCT00360542 (obsolete NCT alias)
Record Dates: First submitted 2006-09-13; First posted 2006-09-15 (Estimated); Results first posted 2014-05-26 (Estimated); Last update posted 2020-02-24 (Actual); Status verified 2020-01

CONDITIONS: Recurrent Breast Carcinoma; Stage III Breast Cancer AJCC v7; Stage IIIA Breast Cancer AJCC v7; Stage IIIB Breast Cancer AJCC v7; Stage IIIC Breast Cancer AJCC v7; Stage IV Breast Cancer AJCC v6 and v7
MeSH Terms: conditions — Breast Neoplasms | interventions — temsirolimus; Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (temsirolimus) (Experimental): Patients receive temsirolimus IV over 30 minutes weekly. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Drug: Temsirolimus

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Temsirolimus — Given IV
  Other Names: CCI-779; CCI-779 Rapamycin Analog; Cell Cycle Inhibitor 779; Rapamycin Analog; Rapamycin Analog CCI-779; Torisel

SUMMARY:
This phase II trial studies how well temsirolimus works in treating patients with breast cancer that has spread to other places in the body. Temsirolimus may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the overall activity (as defined by complete response [CR] + partial response [PR] + stable disease [SD] for >= 24 weeks) of a weekly 25 mg intravenous dose of temsirolimus in patients with locally advanced or metastatic breast cancer.

II. To compare the activity of temsirolimus in patients with locally advanced or metastatic breast cancer whose primary tumors have mutations in the PIK3CA or PTEN gene with those whose tumors do not have a mutation in the PIK3CA gene.

III. To examine correlations between antitumor activity of temsirolimus and alterations in expression of genes in the PI3K pathway in primary tumor biopsy specimens.

OUTLINE:

Patients receive temsirolimus intravenously (IV) over 30 minutes weekly. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed metastatic or recurrent breast cancer not amenable to local therapy (surgery and radiation) (histologic/cytologic confirmation of recurrence preferred, but not required)
* Either the primary or metastatic tumor must be positive for estrogen receptor (>= 1% by immunohistochemical staining) and/or progesterone receptor (>= 1% by immunohistochemical staining) and/or human epidermal growth factor receptor (HER2neu) (3+ immunohistochemical staining or fluorescence in situ hybridization [FISH] positive)
* Patients must have measurable disease; measurable disease is defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as >= 20 mm with conventional techniques or as >= 10 mm with spiral computed tomography (CT) scan
* There are no limitations on the number of prior therapy regimens; however, patients who have had prior exposure to rapamycin or any other mechanistic target of rapamycin (mTOR) inhibitor are excluded from the trial
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* Absolute neutrophil count >= 1,500/uL
* Platelets >= 100,000/uL
* Total bilirubin =< institutional upper limit of normal
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 3 times institutional upper limit of normal
* Creatinine =< 2.0 x normal institutional upper limit of normal
* Cholesterol =< 350 mg/dL (fasting)
* Triglycerides =< 400 mg/dL (fasting)
* Albumin >= 3.3 mg/dL
* Women of child-bearing potential and men must agree to use adequate contraception (barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately; women of child-bearing potential must have a negative pregnancy test prior to treatment on study; breastfeeding should be discontinued if the mother is treated with temsirolimus
* Ability to understand and the willingness to sign a written informed consent document
* Tissue for correlative studies must be available and the subject must agree to use of tissue for these studies

Exclusion Criteria:

* Patients must be off of hormonal agents used for the treatment of breast cancer for one week with the exception that premenopausal women who have been on a gonadotropin-releasing hormone (GnRH) agonist and subsequently progressed may, at the discretion of the treating physician, continue on the GnRH agonist

  * Patients should have recovered from the adverse effects of prior chemotherapy; in general, this will mean that the patient would have been due or overdue for the next dose of the prior regimen: three weeks should have elapsed for a regimen administered once every three weeks, etc
  * Radiotherapy should have been completed
  * Three weeks should have elapsed since prior therapy with monoclonal antibodies
* Patients may not be receiving any other investigational agents or herbal preparations; patients may not be taking corticosteroids except in low doses as replacement for adrenal insufficiency or for short -term (less than 5 days) use for other reasons
* Patients with known brain metastases are not permitted on study unless the metastases have been controlled by prior surgery or radiotherapy, and the patient has been neurologically stable and off of steroids for at least 4 weeks
* Patients cannot be receiving enzyme-inducing antiepileptic drugs (enzyme-inducing antiepileptic drugs [EIAEDs]; e.g., phenytoin, carbamazepine, phenobarbital) nor any other CYP3A4 inducer such as rifampin or St. John's wort, as these may decrease temsirolimus levels; use of agents that potently inhibit CYP3A (and hence may raise temsirolimus levels), such as ketoconazole, is discouraged, but not specifically prohibited; CCI-779 can inhibit CYP2D6, and may decrease metabolism (and increase drug levels) of drugs that are substrates for CYP2D6, such as codeine; the appropriateness of use of such agents is left to physician discretion; if there is any doubt about eligibility based on concomitant medication, the study chair, Dr Fleming, should be contacted; all concomitant medications must be recorded
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, uncontrolled symptomatic cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Human immunodeficiency virus (HIV)-positive patients receiving combination anti-retroviral therapy are excluded from the study
* Patients with known hypersensitivity reactions to macrolide antibiotics (such as erythromycin, clarithromycin, and azithromycin) are not eligible for this trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2006-07-11 (Actual); Primary Completion 2008-06-12 (Actual); Study Completion 2019-12-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gini F Fleming, Principal Investigator — University of Chicago Comprehensive Cancer Center
Locations (2):
- United States (2):
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Washington University School of Medicine, St Louis, Missouri

RESULTS

PARTICIPANT FLOW:
Groups:
- Temsirolimus: Patients receive temsirolimus IV over 30 minutes on days 1, 8, 15, and 22. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Temsirolimus: Given IV
Period: Overall Study
Arm/Group | Temsirolimus
Started | 31
Completed | 27
Not Completed | 4
Not completed — Adverse Event | 3
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Population: Entire study population
Groups:
- Treatment (Temsirolimus): Patients receive temsirolimus IV over 30 minutes on days 1, 8, 15, and 22. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Temsirolimus: Given IV
Arm/Group | Treatment (Temsirolimus)
Number analyzed (Participants) | 31
Age, Continuous [Median (Full Range); unit: years] | 58 [37 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Clinical Benefit Rate (Complete Response, Partial Response, or Stable Disease)
Description: Response evaluation criteria in solid tumors (RECIST) criteria version 1.0 was used for response evaluation. Clinical benefit rate is defined as the proportion of subjects experiencing a complete response (CR), partial response (PR), or stable disease (SD) for at least 24 weeks.
  Evaluation of target lesions: Complete Response (CR)-- Disappearance of all target lesions; Partial Response (PR)-- At least a 30% decrease in the sum of the LD of target lesions, taking as reference the baseline sum LD; Stable Disease (SD)-- Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum LD since the treatment started;
  Evaluation of non-target lesions: Complete Response (CR)-- Disappearance of all non-target lesions and normalization of tumor marker level; Incomplete Response/ Stable Disease (SD)-- Persistence of one or more non-target lesion(s) or/and maintenance of tumor marker level above the normal limits
Time Frame: Up to 24 months
Measure: Number; unit: percentage of participants
Arm/Group | Treatment (Temsirolimus)
Number analyzed (Participants) | 31
percentage of participants | 9.7

ADVERSE EVENTS:
Time Frame: 5 years
Arm/Group | Treatment (Temsirolimus)
Serious Adverse Events (participants affected / at risk) | 9/31
Other Adverse Events (participants affected / at risk) | 16/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Temsirolimus) (N=31)
Abdominal pain (Gastrointestinal disorders) | 2 — A disorder characterized by a sensation of marked discomfort in the abdominal region.
Death NOS (General disorders) | 3 — A cessation of life that cannot be attributed to a CTCAE term associated with Grade 5.
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5 — A disorder characterized by an uncomfortable sensation of difficulty breathing.
Nausea (Gastrointestinal disorders) | 2 — A disorder characterized by a queasy sensation and/or the urge to vomit.
Platelet count decreased (Investigations) | 2 — A finding based on laboratory test results that indicate a decrease in number of platelets in a blood specimen.
Vomiting (Gastrointestinal disorders) | 2 — A disorder characterized by the reflexive act of ejecting the contents of the stomach through the mouth.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Temsirolimus) (N=31)
Alanine aminotransferase increased (Investigations) | 2 — A finding based on laboratory test results that indicate an increase in the level of alanine aminotransferase (ALT or SGPT) in the blood specimen.
Alkaline phosphatase increased (Investigations) | 2 — A finding based on laboratory test results that indicate an increase in the level of alkaline phosphatase in a blood specimen.
Aspartate aminotransferase increased (Investigations) | 2 — A finding based on laboratory test results that indicate an increase in the level of aspartate aminotransferase (AST or SGOT) in a blood specimen.
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 — A disorder characterized by an uncomfortable sensation of difficulty breathing.
Fatigue (General disorders) | 2 — A disorder characterized by a state of generalized weakness with a pronounced inability to summon sufficient energy to accomplish daily activities.
Hyperglycemia (Metabolism and nutrition disorders) | 2 — A disorder characterized by laboratory test results that indicate an elevation in the concentration of blood sugar. It is usually an indication of diabetes mellitus or glucose intolerance.
Hyponatremia (Metabolism and nutrition disorders) | 2 — A disorder characterized by laboratory test results that indicate a low concentration of sodium in the blood.
Hypophosphatemia (Metabolism and nutrition disorders) | 3 — A disorder characterized by laboratory test results that indicate a low concentration of phosphates in the blood.
Lymphocyte count decreased (Investigations) | 7 — A finding based on laboratory test results that indicate a decrease in number of lymphocytes in a blood specimen.
Neutrophil count decreased (Investigations) | 2 — A finding based on laboratory test results that indicate a decrease in number of neutrophils in a blood specimen.
Platelet count decreased (Investigations) | 2 — A finding based on laboratory test results that indicate a decrease in number of platelets in a blood specimen.
White blood cell decreased (Investigations) | 2 — A finding based on laboratory test results that indicate an decrease in number of white blood cells in a blood specimen.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less